CLINICAL TRIAL: NCT02425306
Title: A Trial to Evaluate the Immunogenicity and Safety of a Melanoma Helper Peptide Vaccine Plus Novel Adjuvant Combinations (MEL63)
Brief Title: Safety Study of a Helper Peptide Vaccine Plus Adjuvant Combinations for the Treatment of Melanoma
Acronym: Mel63; CHAMP
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual to part 2 of the study. Accrual to part 1 is complete.
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: Ludwig Institute for Cancer Research (Other); Cancer Research Institute, New York City (Other)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Director, Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17860
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Results first posted 2021-04-29 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Melanoma
Keywords: peptide; vaccine; adjuvant; polyICLC; cyclophosphamide; Montanide ISA-51
MeSH Terms: conditions — Melanoma | interventions — montanide ISA 51; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A:6MHP + Montanide ISA-51 (Experimental): Part 1: 200 mcg of 6MHP emulsified in Montanide ISA-51 adjuvant will be administered on 1, 8, 15, 36, 57 and 78.
  Interventions: Biological: 6MHP; Drug: Montanide ISA-51
- Arm B:6MHP + Montanide ISA-51 + Cyclophosphamide (Experimental): Part 1: 200 mcg of 6MHP emulsified in Montanide ISA-51 adjuvant will be administered on 1, 8, 15, 36, 57 and 78. Cyclophosphamide (50 mg) will be taken orally once a day for 7 days followed by a 7 day rest period. This will be repeated for 5 cycles. Cycles will begin on the following days:
  * Day -6 (Cycle 1)
  * Day 8 (Cycle 2)
  * Day 22 (Cycle 3)
  * Day 36 (Cycle 4)
  * Day 50 (Cycle 5)
  Interventions: Biological: 6MHP; Drug: Montanide ISA-51; Drug: Cyclophosphamide
- Arm C:6MHP + polyICLC + Montanide ISA-51 (Experimental): Part 1: 200 mcg of 6MHP plus 1 mg of polyICLC emulsified in Montanide ISA-51 adjuvant will be administered on 1, 8, 15, 36, 57 and 78.
  Interventions: Biological: 6MHP; Drug: Montanide ISA-51; Drug: polyICLC
- Arm D:6MHP + polyICLC + Montanide ISA-51 + Cyclophosphamide (Experimental): Parts 1 and 2: 200 mcg of 6MHP plus 1 mg of polyICLC emulsified in Montanide ISA-51 adjuvant will be administered on 1, 8, 15, 36, 57 and 78. Cyclophosphamide (50 mg) will be taken orally once a day for 7 days followed by a 7 day rest period. This will be repeated for 5 cycles. Cycles will begin on the following days:
  * Day -6 (Cycle 1)
  * Day 8 (Cycle 2)
  * Day 22 (Cycle 3)
  * Day 36 (Cycle 4)
  * Day 50 (Cycle 5)
  Interventions: Biological: 6MHP; Drug: Montanide ISA-51; Drug: polyICLC; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: 6MHP — 6 melanoma helper vaccine comprised of 6 class II MHC-restricted helper peptides
  Other Names: 6 melanoma helper peptide vaccine
Drug: Montanide ISA-51 — Montanide ISA-51 (Incomplete Freund's Adjuvant), local adjuvant
Drug: polyICLC — polyICLC, local adjuvant
  Arms: Arm C:6MHP + polyICLC + Montanide ISA-51; Arm D:6MHP + polyICLC + Montanide ISA-51 + Cyclophosphamide
Drug: Cyclophosphamide — Cyclophosphamide, systemic adjuvant
  Arms: Arm B:6MHP + Montanide ISA-51 + Cyclophosphamide; Arm D:6MHP + polyICLC + Montanide ISA-51 + Cyclophosphamide

SUMMARY:
This study evaluates whether it is safe to administer a peptide vaccine in combination with different adjuvants. Adjuvants are substances that may boost immune responses vaccines. In this study, the adjuvants are Montanide ISA-51, polyICLC and cyclophosphamide. This study will also evaluate the effects of the combination of the peptide vaccine and the adjuvants on the immune system. The investigators will monitor these effects by performing tests in the laboratory on participants' blood, a lymph node, and tissue from the sites of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 only: Participants with stage IIB, IIC, III, or IV melanoma at original diagnosis or at restaging after recurrence. Patients with high-risk stage IIA melanoma (by DecisionDx Melanoma test, Castle Biosciences, Inc,;Friendswood, TX) also may be eligible. These participants may have had cutaneous, uveal, mucosal primary melanoma, or an unknown primary melanoma. Diagnosis of melanoma must be confirmed by cytological or histological examination. Staging of cutaneous melanoma will be based on version 7 AJCC staging system.
* Part 2 only: Patients with a diagnosis of stage IIIB-IV melanoma with one or more tumor deposits accessible for biopsy and/or excision. These participants may have had cutaneous, uveal, mucosal primary melanoma, or an unknown primary melanoma. Diagnosis of melanoma must be confirmed by cytological or histological examination. Staging of cutaneous melanoma will be based on version 7 AJCC staging system.

Patients must have adequate cutaneous, subcutaneous, soft tissue, or nodal metastases of melanoma readily accessible for biopsy

* Participants will be required to have radiological studies to rule out radiologically evident disease. Required studies include:

  * Chest CT scan,
  * Abdominal and pelvic CT scan, and
  * Head CT scan or MRI
  * PET/CT fusion scan may replace scans of the chest, abdomen, and pelvis.
* Participants who have had brain metastases will be eligible if all of the following are true:

  * Each brain metastasis must have been completely removed by surgery or each unresected brain metastasis must have been treated with stereotactic radiosurgery.
  * There has been no evident growth of any brain metastasis since the most recent treatment.
  * No brain metastasis is > 2 cm in diameter at the time of registration.
  * The most recent surgical resections or gamma-knife therapy for malignant melanoma must have been completed ≥ 1 week and for Part 1, ≤ 6 months prior to registration.
* All participants must have:

  * ECOG performance status of 0 or 1 (Appendix 3)
  * Ability and willingness to give informed consent
* Laboratory parameters as follows:

  * ANC > 1000/mm3
  * Platelets > 100,000/mm3
  * Hgb > 9 g/dL
  * HgbA1c ≤ 7.5%
  * Hepatic:
  * AST and ALT ≤ 2.5 x upper limits of normal (ULN)
  * Bilirubin ≤ 2.5 x ULN (except in patients with Gilbert's disease, where bilirubin to 4x ULN is allowed)
  * Alkaline phosphatase ≤ 2.5 x ULN
  * Renal
  * Creatinine ≤ 1.5 x ULN
  * Serology (within 6 months of study entry)
  * HIV negative
  * Hepatitis C negative (no evidence of active virus)
* Blood is to be collected for HLA typing (Class I and Class II), which will be analyzed as part of the immunologic endpoints, but HLA type will not be an inclusion/exclusion criterion.
* Age 18 years or older at registration.
* Part 1 only: Participants must have at least two intact (undissected) axillary and/or inguinal lymph node basins.
* Part 2 only: Participants must have at least one intact (undissected) axillary and/or inguinal lymph node basin.

Exclusion Criteria:

* Participants who have received the following medications or treatments at any time within 4 weeks of registration:

  * Chemotherapy
  * Interferon (e.g. Intron-A®)
  * Radiation therapy (Stereotactic radiotherapy, such as gamma knife, can be used ≥ 1 week and ≤ 6 months prior to registration)
  * Allergy desensitization injections
  * High doses of systemic corticosteroids, with the following qualifications and exceptions:

    * In patients with adrenal or pituitary insufficiency replacement steroid doses are allowed; however, daily doses of 10 mg or more of prednisone (or equivalent) per day administered parenterally or orally are not allowed in patients with normal adrenal and pituitary function.
    * Inhaled steroids (e.g.: Advair®, Flovent®, Azmacort®) are permitted at low doses (less than 500 mcg fluticasone per day, or equivalent) (76,77).
    * Topical, nasal, and intra-articular corticosteroids are acceptable.
  * Growth factors (e.g. Procrit®, Aranesp®, Neulasta®)
  * Interleukins (e.g. Proleukin®)
  * Any investigational medication
  * Targeted therapies specific for mutated BRAF or for MEK
* Participants who are currently receiving nitrosoureas or who have received this therapy within the preceding 6 weeks
* Participants who are currently receiving a checkpoint molecule blockade therapy, or who have received this therapy within the preceding 12 weeks.
* Participants with known or suspected allergies to any component of the vaccine.
* Participants may not have been vaccinated previously with any of the synthetic peptides included in this protocol. Participants who have received vaccinations containing agents other than the synthetic peptides included in this protocol and have recurred during or after administration of the vaccine will be eligible to enroll 12 weeks following their last vaccination.
* Pregnancy. Female participants of childbearing potential must have a negative pregnancy test (urinary or serum beta-HCG) obtained within 2 weeks prior to registration. Males and females must agree, in the consent form, to use effective birth control methods during the course of vaccination.
* Female participants must not be breastfeeding
* Participants in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol in the opinion of the investigator.
* Participants classified according to the New York Heart Association classification as having Class III or IV heart disease (Appendix 4).
* Participants with uncontrolled diabetes, defined as having a HgbA1c ≥ 7.5%.
* Participants must not have had prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement. Participants with an active autoimmune disorder requiring these therapies are also excluded. The following will not be exclusionary:

  * The presence of laboratory evidence of autoimmune disease (e.g. positive ANA titer) without symptoms
  * Clinical evidence of vitiligo
  * Other forms of depigmenting illness
  * Mild arthritis requiring NSAID medications
* Participants who have another cancer diagnosis, except that the following diagnoses will be allowed:

  * squamous cell cancer of the skin without known metastasis
  * basal cell cancer of the skin without known metastasis
  * carcinoma in situ of the breast (DCIS or LCIS)
  * carcinoma in situ of the cervix
  * any cancer without distant metastasis that has been treated successfully, without evidence of recurrence or metastasis for over 5 years
* Participants with known addiction to alcohol or drugs who are actively taking those agents, or participants with recent (within 1 year) or ongoing illicit IV drug use.
* Body weight < 110 pounds (without clothes) at registration, due to the amount and frequency with which blood will be drawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2018-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L. Slingluff, Jr., MD, Principal Investigator — University of Virginia
Locations (1):
- Cancer Center at the University of Virginia, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open to accrual: May 12, 2015 Close to accrual: June 21, 2018
  Participants all enrolled at an academic medical center.
Groups:
- Arm B:6MHP + Montanide ISA-51 + Cyclophosphamide: Part 1: 200 mcg of 6MHP emulsified in Montanide ISA-51 adjuvant will be administered on 1, 8, 15, 36, 57 and 78. Cyclophosphamide (50 mg) will be taken orally once a day for 7 days followed by a 7 day rest period. This will be repeated for 5 cycles. Cycles will begin on the following days:
  * Day -6 (Cycle 1)
  * Day 8 (Cycle 2)
  * Day 22 (Cycle 3)
  * Day 36 (Cycle 4)
  * Day 50 (Cycle 5)
    6MHP: 6 melanoma helper vaccine comprised of 6 class II MHC-restricted helper peptides
  Montanide ISA-51: Montanide ISA-51 (Incomplete Freund's Adjuvant), local adjuvant
  Cyclophosphamide: Cyclophosphamide, systemic adjuvant
- Arm D:6MHP + polyICLC + Montanide ISA-51 + Cyclophosphamide: Parts 1 and 2: 200 mcg of 6MHP plus 1 mg of polyICLC emulsified in Montanide ISA-51 adjuvant will be administered on 1, 8, 15, 36, 57 and 78. Cyclophosphamide (50 mg) will be taken orally once a day for 7 days followed by a 7 day rest period. This will be repeated for 5 cycles. Cycles will begin on the following days:
  * Day -6 (Cycle 1)
  * Day 8 (Cycle 2)
  * Day 22 (Cycle 3)
  * Day 36 (Cycle 4)
  * Day 50 (Cycle 5)
    6MHP: 6 melanoma helper vaccine comprised of 6 class II MHC-restricted helper peptides
  Montanide ISA-51: Montanide ISA-51 (Incomplete Freund's Adjuvant), local adjuvant
  polyICLC: polyICLC, local adjuvant
  Cyclophosphamide: Cyclophosphamide, systemic adjuvant
Period: Overall Study
Arm/Group | Arm A:6MHP + Montanide ISA-51 | Arm B:6MHP + Montanide ISA-51 + Cyclophosphamide | Arm C:6MHP + polyICLC + Montanide ISA-51 | Arm D:6MHP + polyICLC + Montanide ISA-51 + Cyclophosphamide
Started | 3 | 7 | 6 | 32
Completed | 3 | 6 | 5 | 18
Not Completed | 0 | 1 | 1 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A:6MHP + Montanide ISA-51 | Arm B:6MHP + Montanide ISA-51 + Cyclophosphamide | Arm C:6MHP + polyICLC + Montanide ISA-51 | Arm D:6MHP + polyICLC + Montanide ISA-51 + Cyclophosphamide | Total
Number analyzed (Participants) | 3 | 7 | 6 | 32 | 48
Age, Continuous [Median (Full Range); unit: years] | 48 [45 to 66] | 61 [29 to 79] | 51 [46 to 67] | 59 [30 to 79] | 58 [29 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 11 | 18
  Male | 1 | 4 | 4 | 21 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 7 | 6 | 32 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 7 | 6 | 31 | 47
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 7 | 6 | 32 | 48
AJCC stage (v7) [Count of Participants; unit: Participants] — Each participant was staged according to AJCC version 7 criteria at the time of study enrollment. Risk of death is generally higher for stage III than stage II, and within each stage, risk is higher for stage C than B than A. For those enrolled within 6 months of definitive therapy of the original diagnosis, the stage at diagnoses is used. For those enrolled after a subsequent recurrence or metastasis, the stage at recurrence was used.
  Participants
    AJCC (v7) Stage IIA | 0 | 0 | 0 | 2 | 2
    AJCC (v7) Stage IIB/IIC | 0 | 1 | 1 | 6 | 8
    AJCC (v7) Stage III | 2 | 6 | 5 | 21 | 34
    AJCC (v7) Stage IV | 1 | 0 | 0 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Treatment-related adverse events, by CTCAE v4, Dose-limiting toxicities.
Time Frame: 30 days after administration of the last dose of 6MHP or cyclophosphamide
Population: All 48 participants , including 47 on part 1 and 1 on part 2.
Measure: Number; unit: participants
Arm/Group | Arm A:6MHP + Montanide ISA-51 | Arm B:6MHP + Montanide ISA-51 + Cyclophosphamide | Arm C:6MHP + polyICLC + Montanide ISA-51 | Arm D:6MHP + polyICLC + Montanide ISA-51 + Cyclophosphamide
Number analyzed (Participants) | 3 | 7 | 6 | 32
participants | 0 | 1 | 0 | 2

2. Primary Outcome: Immunogenicity-CD4+ T Cell Responses
Description: CD4+ T cell responses to 6 MHP: durable helper T cell response to 6MHP at 2 or more consecutive timepoints in the PBMC.
Time Frame: through day 85
Population: All ennrolled and treated patients on Parts 1 and 2 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A:6MHP + Montanide ISA-51 | Arm B:6MHP + Montanide ISA-51 + Cyclophosphamide | Arm C:6MHP + polyICLC + Montanide ISA-51 | Arm D:6MHP + polyICLC + Montanide ISA-51 + Cyclophosphamide
Number analyzed (Participants) | 3 | 7 | 6 | 32
Participants | 0 | 2 | 4 | 15

3. Primary Outcome: Immunogenicity-modification of the Tumor Microenvironment (Part 2 Only)
Description: increased infiltration of CD4+ and CD8+ T lymphocytes into melanoma metastases
Time Frame: through day 22
Population: One patient enrolled on Part 2, was on Arm D.
Measure: Number; unit: cells per mm2 of tumor
Arm/Group | Arm A:6MHP + Montanide ISA-51 | Arm B:6MHP + Montanide ISA-51 + Cyclophosphamide | Arm C:6MHP + polyICLC + Montanide ISA-51 | Arm D:6MHP + polyICLC + Montanide ISA-51 + Cyclophosphamide
Number analyzed (Participants) | 0 | 0 | 0 | 1
cells per mm2 of tumor
  CD8 T cells per mm2 in tumor pre-vaccine (day 0) |  |  |  | 401
  CD8 T cells per mm2 in tumor day 22 |  |  |  | 293
  CD4 T cells per mm2 of tumor prevaccine (day 0) |  |  |  | 1202
  CD4 T cells per mm2 tumor day 22 |  |  |  | 1102

4. Secondary Outcome: Immunogenicity-CD8+ T Cell Responses
Description: CD8+ T cell responses to defined melanoma antigens
Time Frame: through day 85
Population: Data were not collected for this endpoint. Funding for this trial has ended.
Arm/Group | Arm A:6MHP + Montanide ISA-51 | Arm B:6MHP + Montanide ISA-51 + Cyclophosphamide | Arm C:6MHP + polyICLC + Montanide ISA-51 | Arm D:6MHP + polyICLC + Montanide ISA-51 + Cyclophosphamide
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through administration of the last dose of 6MHP or mCy, plus 30 days. The scheduled dosing was designed such that the last does of 6MHP vaccine was to be given on day 78 and that the last dose of mCy was to be given on day 57. Thus, for a participant treated on schedule, and to completion, the AE period was 108 days. However, if either or both agents were given for a shorter period (eg held for toxicity), then the time period may be shorter.
Description: The study will be monitored continuously for treatment-related adverse events.
  A DLT is defined as any unexpected adverse event that is possibly, probably or definitely related to treatment and meets the following criteria:
  * ≥ Grade 3
  * ≥ Grade 1 ocular adverse events as defined below
  * ≥ Grade 2 allergic/autoimmune reactions as defined below Exceptions are made for small vaccine site ulceration, and for some transient systemic AEs.
Arm/Group | Arm A:6MHP + Montanide ISA-51 | Arm B:6MHP + Montanide ISA-51 + Cyclophosphamide | Arm C:6MHP + polyICLC + Montanide ISA-51 | Arm D:6MHP + polyICLC + Montanide ISA-51 + Cyclophosphamide
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7 | 0/6 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/7 | 0/6 | 0/32
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 6/6 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A:6MHP + Montanide ISA-51 (N=3) | Arm B:6MHP + Montanide ISA-51 + Cyclophosphamide (N=7) | Arm C:6MHP + polyICLC + Montanide ISA-51 (N=6) | Arm D:6MHP + polyICLC + Montanide ISA-51 + Cyclophosphamide (N=32)
sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant 22 developed septic joint near site of recent trauma, leading to grade 4 sepsis, considered only possibly related to cyclophosphamide but unrelated to the peptides or adjuvants. The patient was taken off study after 2 vaccines.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A:6MHP + Montanide ISA-51 (N=3) | Arm B:6MHP + Montanide ISA-51 + Cyclophosphamide (N=7) | Arm C:6MHP + polyICLC + Montanide ISA-51 (N=6) | Arm D:6MHP + polyICLC + Montanide ISA-51 + Cyclophosphamide (N=32)
Injection site reaction (General disorders) | 3 | 7 | 6 | 32 — Vaccine site local reaction
Skin induration (Skin and subcutaneous tissue disorders) | 3 | 7 | 6 | 32 — Induration at vaccine sites
Fatigue (General disorders) | 2 | 3 | 4 | 20
Nausea (Gastrointestinal disorders) | 0 | 2 | 4 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 6
Headache (Nervous system disorders) | 0 | 2 | 3 | 5
Chills (General disorders) | 0 | 0 | 2 | 7
Flu-like symptoms (General disorders) | 0 | 1 | 1 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 5
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 8 — At sites of vaccines
fever (General disorders) | 0 | 2 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 5
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 4
Mucositis, oral (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Flushing (Vascular disorders) | 1 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT02425306/Prot_SAP_000.pdf